CLINICAL TRIAL: NCT05903716
Title: The Effects of Systemic Isotretinoin Treatment on Adrenal Steroid and Sex Hormones Level in Severe Acne Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2022.464
Record Dates: First submitted 2023-03-26; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Acne Vulgaris
Keywords: Isotretinoin; Adrenal steroid hormones; Sex hormones
MeSH Terms: conditions — Acne Vulgaris | interventions — Thyroid Function Tests; Isotretinoin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — To investigate the17-OH Progesteroone, DHEA, DHEAS, Androstenedione, Aldosterone, Testosterone, Dihydrotestosterone, Estradiol, 17-OH Pregnenolone, Androsterone, Cortisol, Corticosterone, 11-Deoxycortisol, Progesterone, 21-Deoxycortisololone, 11-Deoxycortisolone, Pregnenolone hormones with LCMS/MS technique a 5 ml blood sample was collected from patients.
  To investigate FSH, LH, Prolactin, Estrogen, Testosterone, free testosterone, DHEA-s, SHBG, TSH, T4 hormone levels will be evaluated by ELISA method a 5 ml blood sample was collected from patients. .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe acne vulgaris: 40 female patients aged 14-20 years, who were diagnosed with severe to moderate acne bulgaris and will be treated with isotretinoin.
  Interventions: Diagnostic Test: Hormone; Drug: Isotretinoin
- Healthy control: 40 female patients aged 14-20 years
  Interventions: Diagnostic Test: Hormone

INTERVENTIONS:
Diagnostic Test: Hormone — At baseline 17-OH Progesterone, DHEA, DHEAS, Androstenedione, Aldosterone, Testosterone, Dihydrotestosterone, Estradiol, 17-OH Pregnenolone, Androsterone, Cortisol, Corticosterone, 11-Degesterone, 21, -Deoxycortisol, Pregnenolone, 11-Deoxycorticostreone hormones will be evaluated.In addition, the FSH, LH, Prolactin, Estrogen, Testosterone, free testosterone, DHEA-s, SHBG, TSH, T4 hormone levels of the patients will be evaluated from all patients
Drug: Isotretinoin — İn the 3rd month of isotretinoin treatment, 17-OH Progesterone, DHEA, DHEAS, Androstenedione, Aldosterone, Testosterone, Dihydrotestosterone, Estradiol, 17-OH Pregnenolone, Androsterone, Cortisol, Corticosterone, 11-Degesterone, 21, -Deoxycortisol, Pregnenolone, 11-Deoxycorticostreone hormones will be evaluated.In addition, the FSH, LH, Prolactin, Estrogen, Testosterone, free testosterone, DHEA-s, SHBG, TSH, T4 hormone levels of the patients will be evaluated by ELISA method
  Groups: Severe acne vulgaris

SUMMARY:
Acne vulgaris is a chronic inflammatory skin disease involving the pilosebaceous unit, affecting approximately 95% of adolescents and young adults.

Follicular hyperkeratinization, increased sebum production, androgen hormones and inflammation play a role in the pathogenesis of acne. Androgens (Testosterone, DHEA-S and DHT) play a role in the development of acne, hypertrophy of the sebaceous glands and increased sebum production. Androgen receptors are located in the basal layer of the sebaceous glands keratinocytes and they are located in the outer sheath of the hair follicle. These receptors are responsible for the proliferative action of keratinocytes.

The relationship between androgen hormones and acne in women and prepubertal children is well known. Many studies have shown a strong association between acne and hyperandrogenism in women.

Systemic isotretinoin therapy can be used in patients with severe acne vulgaris who do not respond to topical and oral antibiotic treatments.

In recent studies, it has been shown that systemic isotretinoin used in acne treatment changes many hormones such as GnRH, FSH, LH, Estrogen, Progesterone, Testosterone, TSH, T4 and Prolactin and causes side effects such as menstrual irregularity and hirsutism.

However, data on the effect of oral isotretinoin on adrenal and sex hormones are contradictory.

In this study, it was aimed to evaluate the effect of oral isotretinoin on adrenal steroid and sex hormone levels and to compare it with a healthy control.

Isotretinoin treatment is started in acne vulgaris patients at a dose of 0.5-0.8mg/kg/day. The total cumulative dose is 120 mg/kg.

At baseline and at the 3rd month of isotretinoin treatment, 17-OH Progesterone, DHEA, DHEAS, Androstenedione, Aldosterone, Testosterone, Dihydrotestosterone, Estradiol, 17-OH Pregnenolone, Androsterone, Cortisol, Corticosterone, 11-Degesterone, 21, -Deoxycortisol, Pregnenolone, 11-Deoxycorticostreone hormones will be evaluated with LCMS/MS technique.

In addition, the FSH, LH, Prolactin, Estrogen, Testosterone, free testosterone, DHEA-s, SHBG, TSH, T4 hormone levels of the patients will be evaluated by ELISA method.

In the baseline 2nd, 3rd, 4th and 6th months of the treatment and 3 months after the treatment, the patients' height, weight, body mass index measurements, VAS scoring of patient treatment satisfaction, Global Acne Severity Score, Acne Quality of Life Score, and Modified Ferriman Gallwey Score for hirsutism will be recorded.

The side effects of isotretinoin such as menstrual irregularity, increased hair growth, and cheilitis, dryness of the oral mucosa, skin dryness, dermatitis seen in patients during treatment will be recorded.

*Hormone tests were performed on 2th and 3rd days of menstruation

ELIGIBILITY:
Inclusion Criteria:

* Severe to moderate acne vulgaris
* 14 - 20 Years old
* Female patients

Exclusion Criteria:

* Male patients
* Patients who received vitamin A or hormone therapy in the last 3 months
* Those with adrenal, thyroid, pituitary gland disease
* Those with psychiatric disorders
* History of drug use that causes acneiform eruption (eg, corticosteroids…)
* Acne conglobata and acne fulminans

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who applied to the Dermatology Outpatient Clinic with the diagnosis of severe acne vulgaris and will receive systemic isotrethionine treatment will be evaluated according to the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
FSH Level | Baseline (Before isotretinoin treatment)
  Evaluation FSH levels in Severe Acne Vulgaris patient Before isotretinoin treatment
FSH Level | 3rd month of isotretinoin treatment
  Evaluation FSH levels in after 3 month of isotretinoin treatment
LH Level | Baseline (Before isotretinoin treatment)
  Evaluation LH levels in Severe Acne Vulgaris patient Before isotretinoin treatment
LH Level | 3rd month of isotretinoin treatment
  Evaluation LH levels after 3 month of isotretinoin treatment
Prolactin Level | Baseline (Before isotretinoin treatment)
  Evaluation Prolactin levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Prolactin Level | 3rd month of isotretinoin treatment
  Evaluation Prolactin levels after 3 month of isotretinoin treatment
Estrogen Level | Baseline (Before isotretinoin treatment)
  Evaluation Estrogen levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Estrogen Level | 3rd month of isotretinoin treatment
  Evaluation Estrogen levels after 3 month of isotretinoin treatment
Testosterone Level | Baseline (Before isotretinoin treatment)
  Evaluation Testosterone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Testosterone Level | 3rd month of isotretinoin treatment
  Evaluation Testosterone levels after 3 month of isotretinoin treatment
Free-Testosterone Level | Baseline (Before isotretinoin treatment)
  Evaluation Free-Testosterone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Free-Testosterone Level | 3rd month of isotretinoin treatment
  Evaluation Free-Testosterone levels after 3 month of isotretinoin treatment
DHEA-s Level | Baseline (Before isotretinoin treatment)
  Evaluation DHEA-s levels in Severe Acne Vulgaris patient Before isotretinoin treatment
DHEA-s Level | 3rd month of isotretinoin treatment
  Evaluation DHEA-s levels after 3 month of isotretinoin treatment
SHBG Level | Baseline (Before isotretinoin treatment)
  Evaluation SHBG levels in Severe Acne Vulgaris patient Before isotretinoin treatment
SHBG Level | 3rd month of isotretinoin treatment
  Evaluation SHBG levels after 3 month of isotretinoin treatment
TSH Level | Baseline (Before isotretinoin treatment)
  Evaluation TSH levels in Severe Acne Vulgaris patient Before isotretinoin treatment
TSH Level | 3rd month of isotretinoin treatment
  Evaluation TSH levels iafter 3 month of isotretinoin treatment
T4 Level | Baseline (Before isotretinoin treatment)
  Evaluation T4 levels in Severe Acne Vulgaris patient Before isotretinoin treatment
T4 Level | 3rd month of isotretinoin treatment
  Evaluation T4 levels after 3 month of isotretinoin treatment
17-OH Progesteroone Level | Baseline (Before isotretinoin treatment)
  Evaluation 17-OH Progesteroone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
17-OH Progesteroone Level | 3rd month of isotretinoin treatment
  Evaluation 17-OH Progesteroone after 3 month of isotretinoin treatment
DHEA(LCMS) Level | Baseline (Before isotretinoin treatment)
  Evaluation DHEA(LCMS) levels in Severe Acne Vulgaris patient Before isotretinoin treatment
DHEA(LCMS) Level | 3rd month of isotretinoin treatment
  Evaluation DHEA(LCMS) levels after 3 month of isotretinoin treatment
DHEA-S(LCMS) Level | Baseline (Before isotretinoin treatment)
  Evaluation DHEAS(LCMS) levels in Severe Acne Vulgaris patient Before isotretinoin treatmen
DHEA-S(LCMS) Level | 3rd month of isotretinoin treatment
  Evaluation DHEAS(LCMS) levels after 3 month of isotretinoin treatment
Androstenedione Level | Baseline (Before isotretinoin treatment)
  Evaluation Androstenedione levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Androstenedione Level | 3rd month of isotretinoin treatment
  Evaluation Androstenedione levels after 3 month of isotretinoin treatment
Aldosterone Level | Baseline (Before isotretinoin treatment)
  Evaluation Aldosterone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Aldosterone Level | 3rd month of isotretinoin treatment
  Evaluation Aldosterone levels after 3 month of isotretinoin treatment
Testosterone(LCMS) Level | Baseline (Before isotretinoin treatment)
  Evaluation Testosterone(LCMS) levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Testosterone(LCMS) Level | 3rd month of isotretinoin treatment
  Evaluation Testosterone(LCMS) levels after 3 month of isotretinoin treatment
Dihydrotestosterone Level | Baseline (Before isotretinoin treatment)
  Evaluation Dihydrotestosterone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Dihydrotestosterone Level | 3rd month of isotretinoin treatment
  Evaluation Dihydrotestosterone levels after 3 month of isotretinoin treatment
Estradiol Level | Baseline (Before isotretinoin treatment)
  Evaluation Estradiol levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Estradiol Level | 3rd month of isotretinoin treatment
  Evaluation Estradiol levels after 3 month of isotretinoin treatment
17-OH Pregnenolone Level | Baseline (Before isotretinoin treatment)
  Evaluation 17-OH Pregnenolone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
17-OH Pregnenolone Level | 3rd month of isotretinoin treatment
  Evaluation 17-OH Pregnenolone levels after 3 month of isotretinoin treatment
Androsterone Level | Baseline (Before isotretinoin treatment)
  Evaluation Androsterone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Androsterone Level | 3rd month of isotretinoin treatment
  Evaluation Androsterone levels after 3 month of isotretinoin treatment
Cortisol Level | Baseline (Before isotretinoin treatment)
  Evaluation Cortisol levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Cortisol Level | 3rd month of isotretinoin treatment
  Evaluation Cortisol levels after 3 month of isotretinoin treatment
Corticosterone Level | Baseline (Before isotretinoin treatment)
  Evaluation Corticosterone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Corticosterone Level | 3rd month of isotretinoin treatment
  Evaluation Corticosterone after 3 month of isotretinoin treatment
11-Deoxycortisol Level | Baseline (Before isotretinoin treatment)
  Evaluation 11-Deoxycortisol levels in Severe Acne Vulgaris patient Before isotretinoin treatment
11-Deoxycortisol Level | 3rd month of isotretinoin treatment
  Evaluation 11-Deoxycortisol levels after 3 month of isotretinoin treatment
Progesterone(LCMS) Level | Baseline (Before isotretinoin treatment)
  Evaluation Progesterone(LCMS) levels in Severe Acne Vulgaris patient Before isotretinoin treatment
Progesterone(LCMS) Level | 3rd month of isotretinoin treatment
  Evaluation Progesterone(LCMS) levels after 3 month of isotretinoin treatment
21-Deoxycortisololone Level | Baseline (Before isotretinoin treatment)
  Evaluation 21-Deoxycortisololone levels in Severe Acne Vulgaris patient Before isotretinoin treatment
21-Deoxycortisololone Level | 3rd month of isotretinoin treatment
  Evaluation 21-Deoxycortisololone levels after 3 month of isotretinoin treatment
11-Deoxycortisolone Level | Baseline (Before isotretinoin treatment)
  Evaluation 11-Deoxycortisolone levels in Severe Acne Vulgaris patient Before isotretinoin treatmen
11-Deoxycortisolone Level | 3rd month of isotretinoin treatment
  Evaluation 11-Deoxycortisolone levels after 3 month of isotretinoin treatment
Pregnenolone Level | Baseline (Before isotretinoin treatment)
  Evaluation Pregnenolone levels in Severe Acne Vulgaris patient Before isotretinoin treatmen
Pregnenolone Level | 3rd month of isotretinoin treatment
  Evaluation Pregnenolone levels after 3 month of isotretinoin treatment

SECONDARY OUTCOMES:
Comparison of hormone levels in acne vulgaris patients and healthy group | Baseline
  Comparison of all hormone levels in acne vulgaris patients and healthy group
Menstrual İrregularity | 2. 4. 6. months and 3 month after treatment
  Evaluation of side effects such as menstrual irregularity that can be seen due to isotretinoin
Relationship between Menstrual irregularity and hormone levels | 3rd month of isotretinoin treatment
  Evaluation of the relationship between menstrual irregularity and changes in hormone levels

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine,Department of Dermatology., Istanbul, Turkey (Türkiye)